CLINICAL TRIAL: NCT05808855
Title: Neurological Outcomes Following Carpal Tunnel Decompression: a Comparison of Tissue Adhesive Material and Suture as Wound-closure Techniques
Brief Title: Neurological Outcomes Following Carpal Tunnel Wound-closure Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Vedran Kovacic, Profesor of Medicine, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 500-03/22-01/42
Record Dates: First submitted 2023-02-25; First posted 2023-04-12 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Carpal Tunnel Syndrome Bilateral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin adhesive (Experimental): two-component skin adhesive Glubran Tiss 2®
  Interventions: Procedure: two-component skin adhesive Glubran Tiss 2®
- suture-based wound closure (Active Comparator): suture-based wound closure
  Interventions: Procedure: skin stitched with transcutaneous nylon suture

INTERVENTIONS:
Procedure: two-component skin adhesive Glubran Tiss 2® — After subcutaneous stitches with 4-0 Coated VicrylTM Plus PS-2, 3/8 (Ethicon Inc., USA); a two-component skin adhesive, 0.35 mL of Glubran Tiss 2® (GEM S.r.l., Viareggio, Italy), will be applied in the open wound. Before bandaging, subjects will rest for 20 seconds for a polymerization process.
  Arms: skin adhesive
Procedure: skin stitched with transcutaneous nylon suture — The skin is stitched with transcutaneous nylon sutures (polypropylene-polyethylene monofilament, non-absorbable surgical suture) 4-0
  Arms: suture-based wound closure

SUMMARY:
single-centre randomised prospective trial will conducted at the University Hospital of Split in Croatia. The investigators plan to enrol 100 patients, randomly assigned to suture-based wound closure (n=50) or tissue adhesive-based wound closure (n=50) with two-component skin adhesive Glubran Tiss 2®. The neurological outcomes will assessed postoperatively during the follow-up period at intervals of 2, 6, and 12 weeks respectively.

DETAILED DESCRIPTION:
All surgical procedures will be performed with a tourniquet and local anaesthesia using 2% lidocaine in the palmar soft tissues and carpal tunnel. For all subjects, the standard carpal canal decompression procedure will began withskin incision in the radial half of the palm, followed by carpal ligament transection and cutting. Following primary closure, two different techniques were used depending on the subject's randomization group:

1. The skin will be stitched with transcutaneous nylon sutures (polypropylene-polyethylene monofilament, non-absorbable surgical suture) 4-0.
2. After subcutaneous stitches with 4-0 Coated VicrylTM Plus PS-2, 3/8 ; a two-component skin adhesive, Glubran Tiss 2® will be applied. Each subject will received 0.35 mL of Glubran Tiss® in the open wound, and before bandaging, subjects rested for 20 seconds for a polymerization process.

The neurological outcomes will assessed postoperatively during the follow-up period at intervals of 2, 6, and 12 weeks respectively.

ELIGIBILITY:
Inclusion Criteria: (all of the above)

* age >18 years
* carpal tunnel syndrome
* weakness of thumb abduction
* with atrophy of the thenar
* median nerve conduction impairment estimated by electromyography

Exclusion Criteria: (one or more)

* threatening haemorrhagic complications (patients with peroral anticoagulation and/or antithrombotic therapy)
* previous wrist trauma or surgery on the wrist region
* another aetiology of neuropathy
* previous allergic reactions (with lidocaine, cyanoacrylate, formaldehyde, tapes, or adhesives)
* personal or family history of keloids or hypertrophic scars
* severe general illness with cachexia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
median nerve sensory values measured electromyographic (EMG) | 2 months
  - median nerve latency (msec)
median nerve sensory values measured electromyographic (EMG) | 2 months
  - median nerve sensory conduction velocity (CV) (m/sec)
median nerve sensory values measured electromyographic (EMG) | 2 months
  - median nerve sensory action potential (SAP) amplitude (mcV)

SECONDARY OUTCOMES:
median nerve motoric values measured electromyographic (EMG) | 2 months
  -median nerve motor amplitude (mcV)
Total EMG severity classification | 2 months
  EMG severity will be classified as:
  1. Nerve conduction studies normal
  2. Minimaly abnormal the median nerve sensory latency (<3.5 msec)
  3. Mild, prolonged median sensory latency (<3.5 msec),but normal median DML
  4. Moderate, prolonged median sensory and DML latencies (>4.2 msec)
  5. Severe, absence of median SAP and prolonged or absent median DML.
median nerve motoric values measured electromyographic (EMG) | 2 months
  -median nerve distal motor latency (DML) (msec)
median nerve motoric values measured electromyographic (EMG) | 2 months
  - median nerve motor conduction velocity (m/sec)

CONTACTS AND LOCATIONS:
Locations (2):
- Croatia (2):
  - Surgery Department, Plastic, Reconstructive and Aesthetic Surgery with Burn Care Division, University Hospital of Split, 21000 Croatia, Split
  - University Hospital of Split, 21000 Croatia, Split

IPD SHARING:
Plan to Share IPD: No
Data will be available on request